CLINICAL TRIAL: NCT00021944
Title: Non-Traditional Cardiovascular Risk Factors in Type 2 Diabetes Mellitus - Ancillary to VA Study of Glycemic Control
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 977; R01HL067690 (NIH)
Record Dates: First submitted 2001-08-10; First posted 2001-08-10 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Diabetes Mellitus; Diabetes Mellitus, Non-insulin Dependent; Heart Diseases
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To test whether novel cardiovascular risk factors are related to the presence and development of atherosclerosis and macrovascular events in Type 2 diabetes mellitus and to determine whether intensive glucose lowering therapy will reduce the levels of these cardiovascular risk factors.

DETAILED DESCRIPTION:
BACKGROUND:

A predominant consequence of Type 2 diabetes mellitus is accelerated development of atherosclerosis related conditions. Conventional cardiovascular risk factors only explain a portion of the excess risk for atherosclerosis in this population. This ancillary study uses the study population and framework of the V A Cooperative study of "Glycemic Control and Complications in DM 2". The Cooperative study is a prospective, two-arm, randomized, controlled, multicenter trial to assess the effects of tight glycemic control, achieved through intensification of treatment, on clinical macrovascular and microvascular complications in patients with Type 2 diabetes mellitus who are in poor glycemic control despite pharmacologic therapy. Cooperative study subjects from multiple sites (340 subjects) are participating in the trial.

The study is in response to an initiative "Ancillary Studies in Heart, Lung, and Blood Disease Trials" released by the National Heart, Lung, and Blood Institute in June 2000.

DESIGN NARRATIVE:

This ancillary study examines non traditional risk factors which may contribute to accelerated cardiovascular disease in Type 2 diabetes and the effects of intensive versus standard glycemic management on these risk factors. Specific short-term primary aims include determining the cross-sectional relationship between baseline levels and the presence of atherosclerosis as measured by electron beam computed tomography assessment of coronary artery (CAC) and abdominal aortic calcium (AAC) and the prevalence of clinical macrovascular disease. An estimated 340 Cooperative study subjects from multiple sites will be asked to participate in this additional study. At their baseline visit, subjects will have additional blood and urine collected for a) VLDL, IDL and LDL subfractions b) measures of in vivo oxidative stress (oxidized-phospholipids on plasma LDL, autoantibodies to epitopes of oxidized LDL, F2-isoprostane levels) c) AGE-LDL levels, and d) markers of endothelial activation/injury (PAI-1, VCAM-1 and ICAM-1) and inflammation (C-reactive protein and fibrinogen). Subjects will also have CAC and AAC determined. After enrollment in the study, participants will have measurements of cardiovascular risk factors repeated at six months. Primary and secondary macrovascular endpoints will be identical to those defined in the VA Cooperative study (Primary: myocardial infarction, cardiovascular death, stroke, congestive heart failure, invasive vascular therapy (coronary or peripheral), and amputation due to ischemic gangrene; Secondary: angina pectoris, transient ischemic attacks, and peripheral artery disease). Statistical methods, depending on the specific aim will include categorical age and sex adjusted analyses, t-tests, and multiple regression models. Long-term aims will include evaluating the prospective relationship of these novel cardiovascular risk factors to the progression of atherosclerosis and the development of macrovascular disease in this same population.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reaven — Carl T. Hayden Veteran Affairs Medical Center

REFERENCES:
- [Background] McLaughlin T, Abbasi F, Lamendola C, Liang L, Reaven G, Schaaf P, Reaven P. Differentiation between obesity and insulin resistance in the association with C-reactive protein. Circulation. 2002 Dec 3;106(23):2908-12. doi: 10.1161/01.cir.0000041046.32962.86. PMID 12460870
- [Background] Reaven PD, Thurmond D, Domb A, Gerkin R, Budoff MJ, Goldman S. Comparison of frequency of coronary artery calcium in healthy Hispanic versus non-Hispanic white men by electron beam computed tomography. Am J Cardiol. 2003 Nov 15;92(10):1198-200. doi: 10.1016/j.amjcard.2003.07.030. PMID 14609596
- [Background] Abbasi F, Chu JW, Lamendola C, McLaughlin T, Hayden J, Reaven GM, Reaven PD. Discrimination between obesity and insulin resistance in the relationship with adiponectin. Diabetes. 2004 Mar;53(3):585-90. doi: 10.2337/diabetes.53.3.585. PMID 14988241
- [Background] Reaven PD, Sacks J; Investigators for the VADT. Coronary artery and abdominal aortic calcification are associated with cardiovascular disease in type 2 diabetes. Diabetologia. 2005 Feb;48(2):379-85. doi: 10.1007/s00125-004-1640-z. Epub 2005 Feb 2. PMID 15688207
- [Background] Israelian-Konaraki Z, Reaven PD. Peroxisome proliferator-activated receptor-alpha and atherosclerosis: from basic mechanisms to clinical implications. Cardiology. 2005;103(1):1-9. doi: 10.1159/000081845. Epub 2004 Nov 2. PMID 15528894
- [Background] Reaven PD, Sacks J; Investigators for the Veterans Affairs Cooperative Study of Glycemic Control and Complications in Diabetes Mellitus Type 2. Reduced coronary artery and abdominal aortic calcification in Hispanics with type 2 diabetes. Diabetes Care. 2004 May;27(5):1115-20. doi: 10.2337/diacare.27.5.1115. PMID 15111530